CLINICAL TRIAL: NCT00252980
Title: CANDIS -Targeted Treatment for Cannabis Disorders
Brief Title: CANDIS - Targeted Treatment for Cannabis Disorders
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Technische Universität Dresden (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 01EB0440
Record Dates: First submitted 2005-11-14; First posted 2005-11-15 (Estimated); Last update posted 2007-01-17 (Estimated); Status verified 2007-01

CONDITIONS: Cannabis Use Disorder
Keywords: Cannabis; Dependence; Marijuana; Substance Abuse Treatment; Psychotherapy,
MeSH Terms: conditions — Marijuana Abuse | interventions — Psychotherapy

INTERVENTIONS:
Behavioral: Psychotherapy

SUMMARY:
The purpose of this study is to develop a modular treatment program for cannabis use disorders and the evaluation of the effectiveness in a controlled clinical study.

DETAILED DESCRIPTION:
Background. Cannabis is the most widely used illicit substance in the whole Western world and rates are further rising. Almost 240.000 adult Germans fulfill DSM-IV criteria for cannabis dependence and 140.000 the criteria for cannabis abuse (past 12-month), respectively. Several studies have revealed a considerable degree of unmet needs for intervention and treatment for cannabis disorders, for example in terms of associated physical, mental health, social and legal problems. The epidemiological significance of the problem is contrasted sharply with (1) strongly increasing treatment demand due to cannabis-related problems, (2) the lack of evidence-based interventions (motivational and early treatment) (3) the lack of specific services, and (4) the lack of treatment programs and components with established efficacy. With regard to treatment research there is a marked deficit with only a handful of studies up to date. Only in the US and Australia, some recent effort was undertaken to develop and evaluate cannabis-specific dependence treatment programs in controlled trials with highly selective samples. However, there are currently no 'state of the art' benchmark programs neither in Germany nor in other European countries that are suitable for routine use.

Aims. (1) To develop a modular treatment program (ST/TST) for cannabis use disorders based on treatment packages and components that have been shown to be effective in previous US and Australian trials, and to adapt these material to the needs of our target population. (2) To demonstrate that this modular treatment package, implying motivational enhancement, cognitive-behavioral and psychosocial problem solving components is efficacious in comparison to a delayed treatment control (DTC) group. (3) Additionally, we test whether the targeted standardized treatment (TST) component tailored to address more specifically core problem areas results in superior short term (3-months) outcomes in these core domains as compared to the ST-group.

Method. A randomized controlled intervention study is proposed. A total of 210 participants will be randomly assigned to two, respectively three study conditions: 1. ST (n=70) including motivational enhancement, cognitive-behavioral, and psychosocial problem solving treatment components, 2. TST (n=70), including the same components as the ST but partly individually matched to the specific problem profile of the patient, and (c) a delayed treatment control group (DTC, n=70). Core outcome variables are total quit rates, number of cannabis use in the past 4 weeks, decrease in ASI scores and retention rate. The core hypothesis will be tested in the combined ST/TST group (n=140). The ASI serves for the allocation algorithms in the TST group and serves as outcome measure for the 3rd hypothesis.

The proposed study is innovative and will result in a considerable advancement of our knowledge about effective treatments in cannabis disorders and will inform about the value of targeted individualized allocation.

ELIGIBILITY:
Inclusion Criteria:

* age 16 or older
* lifetime diagnosis of cannabis abuse or cannabis dependence (according to the DSM-IV criteria
* current (4 wks) regular cannabis use (at least 2 days a week)
* persistent history of regular cannabis use of at least 3 years
* informed consent to the study procedures and assessments

Exclusion Criteria:

* current alcohol or any illicit drug dependence syndrome according to DSM-IV other than due to cannabis
* lifetime history of any psychotic disorder
* current severe episode of Major depression
* current panic-agoraphobic disorder (severe)
* severe learning disability, brain damage or pervasive developmental disorder
* currently acute suicidality
* not fluent in german language
* acute signs of intoxication at screening or baseline assessment due to opiates or any type of stimulants, causing cognitive impairments
* currently in treatment for cannabis-related disorders in other services
* current psychotropic medications with sedatives and antipsychotics

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 210
Dates: Start 2006-01; Study Completion 2007-03

PRIMARY OUTCOMES:
- total quit rates, defined as no evidence of cannabis use during the past 4 weeks as evidenced by self report and a negative urine screen; number of times a cannabis product was used in the past 4 weeks
; decrease in ASI total score; retention rate

SECONDARY OUTCOMES:
- number of slips; relapse; abstinence from all legal drugs; number of times of drug use other than cannabis

CONTACTS AND LOCATIONS:
Overall Officials: Eva Hoch, PhD, Principal Investigator — Departement of Clinical Psychology and Psychotherapy, Dresden University of Technology; Hans-Ulrich Wittchen, PhD, Study Director — Departement of Clinical Psychology and Psychotherapy, Dresden University of Technology; Gerhard Bühringer, PhD, Study Director — Departement of Clinical Psychology and Psychotherapy, Dresden University of Technology
Locations (1):
- Department for Clinical Psychology and Psychotherapy; Technical University of Dresden, Dresden, Germany

REFERENCES:
- [Derived] Hoch E, Noack R, Henker J, Pixa A, Hofler M, Behrendt S, Buhringer G, Wittchen HU. Efficacy of a targeted cognitive-behavioral treatment program for cannabis use disorders (CANDIS). Eur Neuropsychopharmacol. 2012 Apr;22(4):267-80. doi: 10.1016/j.euroneuro.2011.07.014. Epub 2011 Aug 24. PMID 21865014
- See also: homepage of the candis-project (for participants) — http://www.candis-projekt.de